CLINICAL TRIAL: NCT04505384
Title: Acute Effects of Left Bundle Branch Pacing Versus Biventricular Pacing for Cardiac Resynchronization Therapy
Brief Title: Acute Effects of LBBP Versus BVP for CRT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Shanghai Zhongshan Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ZS-LBBPvsBVP
Record Dates: First submitted 2020-07-31; First posted 2020-08-10 (Actual); Last update posted 2022-01-20 (Actual); Status verified 2022-01

CONDITIONS: Heart Failure; Cardiac Pacing, Artificial; Cardiac Resynchronization Therapy
MeSH Terms: conditions — Heart Failure | interventions — Cardiac Resynchronization Therapy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Left bundle branch pacing (Experimental): Left bundle branch pacing
  Interventions: Procedure: left bundle branch pacing
- Biventricular pacing (Active Comparator): Biventricular pacing
  Interventions: Procedure: biventricular pacing

INTERVENTIONS:
Procedure: left bundle branch pacing — left bundle branch pacing
  Arms: Left bundle branch pacing
Procedure: biventricular pacing — biventricular pacing
  Arms: Biventricular pacing

SUMMARY:
The study was designed to compare the acute effects of left bundle branch pacing (LBBP) with biventricular pacing (BVP) in patients with left ventricular ejection fraction (LVEF) <=35% with left bundle branch block (LBBB).

DETAILED DESCRIPTION:
The metrics include electrocardiographic, echocardiographic and hemodynamic parameters to evaluate and compare LBBP with BVP for resynchronization therapy in patients with heart failure and LBBB.

ELIGIBILITY:
Inclusion Criteria:

* NYHA class II-IV;
* LVEF <=35%;
* LBBB with QRS duration >=130ms.

Exclusion Criteria:

* moderate-to-severe aortic stenosis;
* frequent premature ventricular complexes;
* signiﬁcant peripheral vascular disease.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2020-09-01 (Actual); Primary Completion 2021-09-30 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
Hemodynamic parameter LV dP/dt(max) | 1 hour
  LV dP/dt(max) will be obtained during implant procedure.

SECONDARY OUTCOMES:
Electrical synchrony parameters including QRS duration and QRS area | 0.5 hour
  Acquired from EP system during procedure
Mechanical parameters including Ts-SD and IVMD | 0.5 hour
  Acquired by an echocardiologist during procedure

CONTACTS AND LOCATIONS:
Overall Officials: Yangang Su, MD, Study Chair — Shanghai Zhongshan Hospital
Locations (1):
- 180 Fenglin Road, Shanghai, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Liang Y, Wang J, Gong X, Lu H, Yu Z, Zhang L, Li M, Pan L, Chen X, Cui J, Zhang W, Li R, Zhou X, Huang W, Su Y, Ge J. Left Bundle Branch Pacing Versus Biventricular Pacing for Acute Cardiac Resynchronization in Patients With Heart Failure. Circ Arrhythm Electrophysiol. 2022 Nov;15(11):e011181. doi: 10.1161/CIRCEP.122.011181. Epub 2022 Oct 28. PMID 36306335